CLINICAL TRIAL: NCT00851617
Title: Is Threshold IMT Useful To Accelerate Weaning From Mechanical Ventilation?
Brief Title: Does Threshold IMT Influence Weaning?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Federal University of Rio Grande do Sul, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 04-391
Record Dates: First submitted 2009-02-09; First posted 2009-02-26 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-02

CONDITIONS: Critical Care; Mechanical Ventilation
Keywords: Mechanical ventilator weaning; Respiratory Muscle Training; Ventilator dependent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMT Group (Experimental): The IMT group was trained using the threshold IMT device with a 40% MIP load. Each training session consisted of 5 sets with 10 breaths, twice a day
  Interventions: Device: Threshold® IMT
- Control Group (No Intervention): Patients were evaluated until weaning without interventions

INTERVENTIONS:
Device: Threshold® IMT — The IMT group was trained using the threshold IMT device with a 40% MIP load. Each training session consisted of 5 sets with 10 breaths, twice a day
  Arms: IMT Group

SUMMARY:
Patients under threshold IMT show better conditions to weaning from mechanical ventilation than the control group.

DETAILED DESCRIPTION:
* After at least 48 hours on CMV, the patients in PSV were randomized into two groups: control group and IMT group.
* Before each protocol session, the cardiorespiratory variables such as f, HR, MAP and SpO2, as well as the support ventilatory variables such as PSV, PEEP, FiO2 and trigger sensitivity, were recorded.
* After collecting the first records, the patients were placed in a 45º Fowler position, and variables MIP and MEP were collected with a unidirectional valve, as well as f, VE, Vt and f/Vt.
* The IMT group was trained using the threshold IMT device with a 40% MIP load. Each training session consisted of 5 sets with 10 breaths, twice a day. Supplementary oxygen was added if necessary during the protocol. The training was cancelled in the presence of tachyarrhythmia, reduction of SpO2 under 85% and in the presence of fatigue signs or respiratory dysfunction. In this case, the patients returned to MV. All cardiorespiratory variables (f, HR, MAP and SpO2) were recorded again one minute after the end of the protocol. The same data were recorded in the control group before and after the protocol, but the patients were not trained with the threshold IMT device.
* All patients were followed up until weaning. During this period, laboratory tests were recorded, such as: potassium, sodium and magnesium as well as arterial gasometry, calculating the partial pressure of arterial oxygen/fraction of inspired oxygen (PaO2/FiO2) ratio.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study were under MV for more than 48 hours of CMV and ventilated with pressure support ventilation (PSV) between 12 and 15 cmH2O, with positive end-expiratory pressure (PEEP) between 5 and 7 cmH2O, hemodynamically stable without vasoactive drugs (dopamine, dobutamine or norepinephrine) or sedative agents.

Exclusion Criteria:

* This study excluded hypotensive patients (systolic blood pressure < 100 mmHg or mean blood pressure < 70 mmHg), severe intracranial disease and sensory reduction, barotrauma, tracheotomy, neuromuscular disease and the use of vasoactive drugs or sedatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-08; Primary Completion 2005-03 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Weaning Acceleration | Time weaning measured in hours

SECONDARY OUTCOMES:
Strenght and ventilatory variables | Time weaning measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Vieira, PhD, Principal Investigator — Federal University of Rio Grande do Sul, Hospital de Clínicas de Porto Alegre
Locations (1):
- Federal University of Rio Grande do Sul, Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil